CLINICAL TRIAL: NCT04591834
Title: A Prospective, Observational Study of Pediatric Patients With Neuronopathic Forms of MPS II (Hunter Syndrome)
Brief Title: Mucopolysaccharidosis Type II Observational
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor decision
Sponsor: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RGX-121-9101
Record Dates: First submitted 2020-09-23; First posted 2020-10-19 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Mucopolysaccharidosis II
Keywords: MPS II; Gene Therapy; Hunter
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: No Intervention
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — An observational study in subjects with the severe form of MPS II.

SUMMARY:
This is an observational study planned to document prospectively disease manifestation and neurocognitive course in pediatric patients with a clinical presentation consistent with neuronopathic ("severe") MPS II undergoing current standard of care and/or intrathecal Elaprase® for their condition. Some patients may be offered the opportunity to screen for a gene therapy study conducted by the same sponsor.

DETAILED DESCRIPTION:
MPS II is a rare X-linked recessive genetic disease caused by mutations in the iduronate-2-sulfatase gene (IDS). Enzyme replacement therapy (ERT) with recombinant idursulfase (ELAPRASE®) is the only approved product for the treatment of Hunter syndrome; however, ERT as currently administered does not cross the blood brain barrier and is therefore unable to address the unmet need in MPS II patients with CNS (neurocognition and behavior) involvement. This is an observational study to document prospectively disease manifestation and neurocognitive course in pediatric patients with a clinical presentation consistent with neuronopathic ("severe") MPS II undergoing current standard of care for their condition. Approximately forty pediatric subjects who have severe MPS II will be enrolled. Changes in neurodevelopmental parameters of cognitive, behavioral, and adaptive function over time will be the primary focus for a duration of 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Meets any of the following criteria:

   1. Has a clinical diagnosis of severe MPS II and has a documented mutation in IDS, OR
   2. Has a relative clinically diagnosed with severe MPS II who has the same IDS mutation as the subject, OR
   3. Has documented mutation(s) in IDS that in the opinion of the investigator is known to result in a neuronopathic phenotype
2. Has sufficient communication capacity to complete the required protocol testing

Patient's legal guardian must be willing and able to provide written, signed informed consent.

Exclusion Criteria:

1. Has had prior treatment with an AAV-based gene therapy product
2. Is currently participating in a clinical trial of an investigational product for the treatment of MPS II with the exception of IT ELAPRASE trials; no investigational product may be taken starting 30 days or 5 half-lives of the investigational product prior to signing the ICF, whichever is longer

Ages: 1 Month to 8 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Up to 40 subjects ages 1 month to 8 years of age who have documented neurocognitive deficits due to MPS II or who have a genotype and family history consistent with an inherited form of severe MPS II will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Changes in neurodevelopmental parameters of cognitive function over time | 104 weeks
  Bayley Scales of Infant and Toddler Development Third Edition (BSID-III)
Changes in neurodevelopmental parameters of cognitive function over time | 104 weeks
  Mullen Scales of Early Learning (MSEL) Visual Reception Domain
Changes in neurodevelopmental parameters of adaptive behavior function over time | 104 weeks
  Vineland Adaptive Behavior Scales Second Edition (VABS-II)

SECONDARY OUTCOMES:
Changes in disease-specific biomarkers over time | 104 weeks
  I2S activity
Changes in disease-specific biomarkers over time | 104 weeks
  GAGs
Changes in quality of life | 104 weeks
  PedsQL
Changes in quality of life | 104 weeks
  ADL
Changes in Caregiver reported outcome | 104 weeks
  Family Burden of Illness Survey
Changes in sleep | 104 weeks
  SDSC

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - University of California San Francisco, Benioff Children's Hospital, Oakland, California
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- McGill University Health Center, Montreal, Quebec, Canada